CLINICAL TRIAL: NCT06708923
Title: Evaluation of Acupuncture's Effectiveness on Pregnancy Outcomes in Women with Recurrent Implantation Failure RIF: a Large Cohort Study
Acronym: AcupunctureRIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Thi Thanh Thuy Tran, MD, Infertility Specialist, Department of Infertility, Hung Vuong Hospital, Hung Vuong Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS/HV/24/36
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Infertility (IVF Patients); Acupuncture
Keywords: Recurrent Implantation Failure (RIF); Acupuncture; In Vitro Fertilization (IVF)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: This study employs an Observational Retrospective Cohort Design to investigate the impact of acupuncture on pregnancy outcomes in patients diagnosed with recurrent implantation failure (RIF) undergoing frozen embryo transfer (FET) cycles.
  Participants are categorized into two cohorts:
  Acupuncture Cohort: Patients who received acupuncture treatments before and after embryo transfer during their IVF cycle.
  Non-Acupuncture Cohort: Patients who did not receive acupuncture during their IVF cycle.
  The study analyzes historical medical records to compare key clinical outcomes between the two cohorts, including clinical pregnancy rate (CPR), ongoing pregnancy rate (OPR), and live birth rate (LBR).
  No experimental interventions are conducted during the study period, as it relies on previously collected data. Statistical methods are applied to adjust for confounding variables such as age, BMI, and number of prior failed cycles to ensure accurate comparisons and reliable conclusions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IVF with Acupuncture Group: Patients undergoing IVF cycles with acupuncture performed before and aft (Experimental): IVF with Acupuncture Group:
  This group includes patients who underwent IVF cycles with acupuncture performed at two key time points:
  Before Embryo Transfer: Acupuncture was administered 25 minutes prior to transfer at specific acupoints (e.g., Baihui, Guanyuan, Sanyinjiao) to enhance endometrial receptivity and reduce stress.
  After Embryo Transfer: A second acupuncture session was conducted immediately following the transfer at additional acupoints (e.g., Zusanli, Taichong) to support implantation and relaxation.
  IVF without Acupuncture Group:
  This group includes patients who underwent IVF cycles without any acupuncture treatment. Their IVF procedures followed standard clinical protocols for frozen embryo transfer (FET), including hormonal preparation of the endometrium and embryo transfer, without any complementary therapies.
  The study retrospectively compares clinical outcomes, including clinical pregnancy rate (CPR), ongoing pregnancy rate (OPR), and live birth rate (LBR), betwee
  Interventions: Procedure: Intervention Name: Acupuncture Therapy Before and After Embryo Transfer Description: The intervention involves acupuncture therapy performed at two key time points during the IVF cycle: 25 minutes be

INTERVENTIONS:
Procedure: Intervention Name: Acupuncture Therapy Before and After Embryo Transfer Description: The intervention involves acupuncture therapy performed at two key time points during the IVF cycle: 25 minutes be — Acupuncture Therapy Before and After Embryo Transfer
  This intervention consists of acupuncture sessions designed to support implantation and improve pregnancy outcomes during frozen embryo transfer (FET) cycles.
  Procedure:
  Acupuncture is performed using sterile, single-use needles by certified practitioners trained in reproductive health.
  Sessions occur at two critical time points:
  Before Embryo Transfer: A 25-minute session targeting acupoints such as Baihui (DU20), Guanyuan (CV4), and Sanyinjiao (SP6) to enhance endometrial receptivity and reduce stress.
  After Embryo Transfer: A second 25-minute session targeting acupoints such as Zusanli (ST36) and Taichong (LR3) to promote implantation and relaxation.
  Purpose:
  Improve uterine blood flow and receptivity. Regulate hormonal balance to optimize the implantation environment. Reduce psychological stress associated with IVF procedures. This intervention is compared retrospectively to standard IVF protocols without acupuncture to asses

SUMMARY:
Title: Evaluating the Effectiveness of Acupuncture on Pregnancy Outcomes in Recurrent Implantation Failure (RIF) Patients Undergoing In Vitro Fertilization (IVF): A Large Cohort Study

Objective:

This study aims to assess the efficacy of acupuncture in improving pregnancy outcomes, including clinical pregnancy rate (CPR), ongoing pregnancy rate (OPR), and live birth rate (LBR), in patients who have experienced recurrent implantation failure (RIF) during frozen embryo transfer (FET) cycles.

Background:

Recurrent implantation failure (RIF) is a significant challenge in assisted reproductive technologies (ART), affecting approximately 15% of IVF patients. The causes of RIF include uterine factors, embryo quality issues, and immune dysfunctions. Acupuncture, a traditional Chinese medical practice, has gained interest as an adjunctive treatment in IVF, potentially enhancing uterine blood flow, regulating hormones, and alleviating stress. While previous studies suggest a positive impact of acupuncture on IVF outcomes, its role in patients with RIF remains unclear, particularly in Vietnam, where its integration into modern fertility treatments is emerging.

Methods:

Design: Retrospective cohort study. Setting: IVF Department, Hung Vuong Hospital, Ho Chi Minh City. Participants: 1,969 IVF cycles from RIF-diagnosed patients between January 2019 and December 2023, divided into two groups: those who received acupuncture and those who did not.

Interventions:

Acupuncture sessions were performed 25 minutes before and after embryo transfer, targeting specific acupoints (e.g., Baihui, Guanyuan, Sanyinjiao).

Standardized hormonal protocols (HRT-E+P) and embryology practices were applied uniformly across all participants.

Outcome Measures: CPR, OPR, LBR, biochemical pregnancy rates, and miscarriage rates were analyzed.

Statistical Analysis:

Descriptive statistics summarized baseline characteristics. Logistic regression was used to evaluate the association between acupuncture and pregnancy outcomes, adjusting for potential confounders such as age, BMI, and number of prior failed cycles.

Results (Preliminary):

The study hypothesizes that patients receiving acupuncture will demonstrate improved CPR, OPR, and LBR compared to non-acupuncture counterparts. Previous research has suggested a trend toward higher clinical pregnancy rates with acupuncture, but statistical significance and the mechanisms behind these effects require further exploration.

Ethical Considerations:

Patient data were anonymized, and the study was approved by the institutional ethics committee. Participation was voluntary, with informed consent obtained prior to treatment.

Conclusions:

This research seeks to provide robust evidence on the integration of acupuncture into fertility treatment protocols for RIF patients, addressing a critical gap in both global and Vietnamese reproductive healthcare. If proven effective, acupuncture could become a valuable complementary therapy in enhancing IVF success rates.

This study represents a crucial step toward combining traditional and modern medical practices to improve reproductive outcomes.

DETAILED DESCRIPTION:
Study Title: Evaluating the Effectiveness of Acupuncture on Pregnancy Outcomes in Recurrent Implantation Failure (RIF) Patients Undergoing In Vitro Fertilization (IVF): A Large Cohort Study

Background:

Recurrent implantation failure (RIF) is a complex condition that poses significant challenges to the success of assisted reproductive technology (ART). Defined by the European Society of Human Reproduction and Embryology (ESHRE), RIF occurs when a clinical pregnancy is not achieved after the transfer of good-quality embryos in multiple IVF cycles. Causes include embryo quality, uterine abnormalities, immunological factors, and hormonal imbalances. The psychological and physical stress associated with repeated failures further complicates treatment.

Acupuncture, a traditional Chinese medicine practice, has been used for over 3,000 years to treat various conditions. In the context of infertility, acupuncture is believed to enhance uterine blood flow, regulate endocrine function, and reduce patient stress, thus creating a favorable environment for implantation. While prior studies have suggested that acupuncture may improve IVF outcomes, evidence specific to patients with RIF remains limited, particularly in Vietnam, where it has been integrated into modern reproductive medicine only recently.

Objective:

To investigate the impact of acupuncture on pregnancy outcomes, including clinical pregnancy rate (CPR), ongoing pregnancy rate (OPR), and live birth rate (LBR), in patients with RIF undergoing frozen embryo transfer (FET) cycles.

Study Design:

This is a retrospective cohort study conducted at the IVF Department of Hung Vuong Hospital, a leading center for reproductive medicine in Ho Chi Minh City, Vietnam.

Participants:

The study includes 1,969 IVF cycles performed between January 2019 and December 2023 on patients diagnosed with RIF. Patients were categorized into two groups based on whether they received acupuncture during their treatment cycles.

Inclusion Criteria:

Women diagnosed with RIF, defined as the absence of a clinical pregnancy after three or more embryo transfers using good-quality embryos.

At least one viable frozen embryo available for transfer. Endometrial preparation using hormone replacement therapy (HRT-E+P). Written consent from both partners for participation in IVF treatment.

Exclusion Criteria:

Untreated uterine anomalies (e.g., septate uterus). Preimplantation genetic testing (PGT) cycles. Egg or sperm donation. Unmanaged endocrine disorders (e.g., hyperthyroidism, diabetes). Patients without complete medical records or those who did not consent to the use of their data.

Intervention:

Acupuncture was performed at two critical time points during the FET cycle:

Before Embryo Transfer: A session lasting 25 minutes, targeting acupoints such as Baihui (DU20), Guanyuan (CV4), and Sanyinjiao (SP6), aimed at improving uterine receptivity and reducing stress.

After Embryo Transfer: Another 25-minute session targeting points including Zusanli (ST36) and Taichong (LR3), designed to enhance implantation and maintain relaxation.

Standardized acupuncture protocols were developed based on evidence from global and local studies, ensuring consistency in treatment.

Outcome Measures:

Primary Outcomes:

Clinical pregnancy rate (CPR): Presence of a gestational sac on ultrasound. Ongoing pregnancy rate (OPR): Pregnancy sustained beyond 12 weeks. Live birth rate (LBR): Birth of a viable infant.

Secondary Outcomes:

Biochemical pregnancy rate: Positive beta-hCG levels. Miscarriage rates: Early and late pregnancy losses.

Methodology:

Data Collection: Clinical data were extracted from electronic medical records. Information on patient demographics, IVF history, embryo quality, and acupuncture details were recorded.

Acupuncture Protocol: Acupuncture sessions were performed using sterile, single-use needles by certified practitioners trained in reproductive health.

Data Analysis: Statistical analyses were conducted using Stata 14. Logistic regression models adjusted for confounders, including age, BMI, and number of prior failed cycles, were used to evaluate associations between acupuncture and pregnancy outcomes.

Statistical Analysis Plan:

Descriptive statistics summarized baseline characteristics. Chi-square tests and Fisher's exact tests compared pregnancy outcomes between groups.

Logistic regression analysis adjusted for confounding variables, with results reported as odds ratios (OR) and 95% confidence intervals (CI).

Ethical Considerations:

The study was approved by the institutional ethics committee of Hung Vuong Hospital. All participants provided written informed consent for their data to be used in the study. Data were anonymized to ensure confidentiality.

Significance:

This study aims to provide robust evidence regarding the integration of acupuncture into fertility treatments for patients with RIF. By evaluating its impact on various pregnancy outcomes, the study seeks to address a critical gap in both local and global reproductive healthcare. Findings could inform clinical guidelines and promote a multidisciplinary approach combining traditional and modern medicine to improve IVF success rates.

Potential Impact:

If successful, this study could:

Validate acupuncture as an effective adjunctive therapy for RIF patients. Encourage the adoption of acupuncture in reproductive medicine, enhancing holistic patient care.

Provide insights into optimal acupuncture protocols for maximizing IVF success. This research represents a significant step in bridging traditional medicine with cutting-edge reproductive technologies, offering renewed hope to couples facing infertility challenges.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with recurrent implantation failure (RIF), defined as the absence of clinical pregnancy after at least three transfers of good-quality embryos.
2. Patients undergoing frozen embryo transfer (FET) cycles with at least one viable frozen embryo.
3. Endometrial preparation using hormone replacement therapy (HRT-E+P).
4. Complete consent form signed by both partners and the attending physician, as per IVF protocol at Hung Vuong Hospital.
5. Availability of complete clinical and embryological records from January 2019 to December 2023.

Exclusion Criteria:

1. Structural uterine abnormalities, including untreated septate uterus or uterine malformations.
2. Patients undergoing preimplantation genetic testing (PGT) cycles.
3. Use of donor eggs or sperm.
4. Presence of untreated endocrine disorders, including but not limited to hyperthyroidism, hypothyroidism, diabetes, and hypertension.
5. Patients lacking consent for data usage in the study or incomplete clinical records.

Criteria for Recurrent Implantation Failure (RIF)

Definition:

According to the European Society of Human Reproduction and Embryology (ESHRE), recurrent implantation failure (RIF) is defined as the inability to achieve a clinical pregnancy after transferring good-quality embryos across multiple in vitro fertilization (IVF) cycles.

Criteria for RIF Diagnosis:

Number of Transfers: Failure to achieve pregnancy after at least three embryo transfers (fresh or frozen), with a minimum of 1-2 good-quality embryos transferred each time.

Total Number of Embryos: Alternatively, RIF can be defined as failure to achieve pregnancy after transferring at least four good-quality embryos in total.

Possible Causes:

RIF can result from factors related to the embryo, uterus, or other conditions, such as:

Embryo quality issues (e.g., genetic abnormalities or poor development). Uterine abnormalities (e.g., insufficient endometrial thickness or structural anomalies).

Immunological or hematological factors affecting implantation. These criteria guide the identification of patients who may benefit from further investigation or specialized treatments, such as those evaluated in this study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1969 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate (CPR) | 6-8 weeks post-embryo transfer.
  The proportion of participants achieving a clinical pregnancy, defined as the presence of a gestational sac observed via ultrasound after frozen embryo transfer (FET).

SECONDARY OUTCOMES:
Ongoing Pregnancy Rate (OPR) | 12 weeks post-embryo transfer.
  The proportion of participants with a pregnancy that continues beyond the first trimester (12 weeks), confirmed by ultrasound. This measures the sustainability of pregnancy following frozen embryo transfer (FET).
Live Birth Rate (LBR) | Approximately 9 months post-embryo transfer.
  The proportion of participants delivering a live infant after IVF treatment. This is the ultimate indicator of treatment success for both the acupuncture and non-acupuncture groups.

CONTACTS AND LOCATIONS:
Overall Officials: PHUONG HUY TRAN, MSc, Principal Investigator — IVF Hung Vuong
Locations (1):
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No